CLINICAL TRIAL: NCT02815605
Title: Risk Factors, Management and Complications of Severe Post-partum Hemorrhage: A Retrospective Analysis in a Single Tertiary Referral Center
Brief Title: Risk Factors, Management and Complications of Severe Post-partum Hemorrhage
Acronym: PPH-REG
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ETL R16092
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Post-partum Hemorrhage; Blood Transfusion
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of severe post-partum hemorrhage has been increasing in developed countries. The reason for this is at least partially unknown. Surgical techniques, holistic treatment protocols and strategies in blood product administration may have changed patient outcome and, for example the incidence of transfusion related side effects. A retrospective analysis of the whole cohort of parturients in 2009-2015 in Tampere University Hospital will be made to assess the risk factors for severe PPH (ie. estimated blood loss more than 1500ml during delivery) and examine the possible change in blood transfusion strategies and its effect on bleeding (for example, implementation of massive transfusion protocol, amount of blood products used, effect of red blood cell:fresh-frozen plasma ratio, use of pharmacological agents for coagulation management, introduction of new angiological and surgical techniques etc.) and complications, laboratory parameters and patient outcome.

DETAILED DESCRIPTION:
Post-partum haemorrhage (PPH) still remains one of leading causes of morbidity in the obstetric population and a recent report from the United Kingdom revealed that hemorrhage is the sixth most important direct cause of maternal mortality. During labor, the blood flow in the uterus increases and obstetric hemorrhage may quickly turn to massive bleeding requiring massive transfusion of allogeneic blood products. Although introduction of massive transfusion protocols (MTP) may have improved survival in trauma patients, administration of allogeneic blood products, although life-saving, is also associated with considerable side effects. That is why a stepwise progressive approach and implementation of treatment protocols describing the timely use of different pharmacological agents and surgical or radiological interventions are called for. Risk factors for blood transfusion (as a surrogate marker for PPH) at delivery in Finland have been recently studied , and the results seem to be in consonance with reports from several developed countries, which demonstrate a marked increase in incidence of PPH. However, the causes for the increase in postpartum hemorrhage remain at least partly unclear. Also, complication rates of blood transfusion and other adverse outcomes in the treatment of an obstetric patient with severe bleeding are not very recently studied (19). Identification of PPH risk factors, change in transfusion strategies and surgical techniques and implementation of holistic treatment protocols may have had an effect on the complication rate, costs and total amount of blood product usage and bleeding, but to investigators' knowledge, these are underreported in current studies.That is why it seems justified to examine a cohort of parturients with severe PPH under a long time span to find out whether the change in practice is reflected in patients' outcome.

From 2009 to December 2015, all patients having a marked post-partum hemorrhage (estimated blood loss 1500ml) will be tracked from Tampere University hospital's computerized perinatal database (iPana). Approximate number of patients is 900: according to the database, the incidence of severe PPH in our hospital is 130-160/year. General patient characteristics will be recorded: age, weight, height, parity, gestational age, previous deliveries and cesarean sections, chronic diseases, complications and medication during pregnancy. The mode of delivery, labour characteristics (duration, interval between PROM and delivery, chorioamnionitis), use of uterotonic agents and diagnoses of obstetric disease will be recorded (e.g. placental abnormalities). Laboratory parameters during treatment of PPH will be collected: a baseline aPTT, PT (INR), Fibrinogen concentration, ATIII, Hb, platelet count and respective (lowest) values during treatment of PPH and blood gas analysis information, especially lowest base excess and lactate and lowest ca-ion. Other possible factors affecting hemostasis such as body temperature, hemodynamic parameters during resuscitation and surgical treatment will be searched from medical records. Total amount of bleeding and allogeneic blood products, fibrinogen concentrate, prothrombin complex concentrate, FXIII and recombinant factor VII consumption will be recorded as primary end points. As secondary endpoints, the number of emergency hysterectomies, intensive care admissions, transfusion-related side effects and thromboembolic complications will be studied and recorded up to 30 days after delivery.

The investigators' aim is to identify risk factors for severe PPH (ie. estimated blood loss more than 1500ml during delivery) and examine the possible change in blood transfusion strategies and its effect on bleeding (for example, implementation of massive transfusion protocol, amount of blood products used, effect of red blood cell:fresh-frozen plasma ratio, use of pharmacological agents for coagulation management, introduction of new angiological and surgical techniques etc.) and complications, laboratory parameters and patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18,
* Severe post-partum hemorrhage ie. active bleeding more than 1500ml within 24 hours after vaginal delivery or cesarean section.

Exclusion Criteria:

* Known hemophilia,
* Severe (type 2 and forth) von Willebrandt's disease or thrombasthenia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All parturients in 2009-2015 in Tampere University Hospital with severe post-partum hemorrhage ie. active bleeding more than 1500ml within 24 hours after vaginal delivery or cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Total amount of bleeding | 2009-2015
  in millilitres
Blood component usage | 2009-2015
  Number of red cell, Octaplas (R) and thrombocyte units administered
Use of procoagulant medication | 2009-2015
  Amount of fibrinogen concentrate, prothrombin complex concentrate, FXIII and recombinant factor VII administered

SECONDARY OUTCOMES:
Number of emergency hysterectomies | 2009-2015
Number of Intensive care admissions | 2009-2015
Transfusion-related side effects and thromboembolic complications | 2009-2015
  Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kuitunen, MD, PhD, Study Director — Tampere University Hospital; Samuli Jokinen, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided